CLINICAL TRIAL: NCT00771017
Title: A Randomized, Phase II Trial of Brief Androgen-Ablation Combined With Cell-based CG1940/CG8711 Immunotherapy For Prostate Cancer in Patients With Non-Metastatic, Biochemically Relapsed Prostate Cancer
Brief Title: Androgen Ablation Therapy With or Without Vaccine Therapy in Treating Patients With Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000616570; ECOG-E3806
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage II prostate cancer; stage III prostate cancer; stage I prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Goserelin; Leuprolide

ARMS (2):
- Arm I (Active Comparator): Patients receive oral bicalutamide once daily on days 1-28. Patients also receive luteinizing-hormone releasing-hormone (LHRH) agonist treatment comprising leuprolide acetate or goserelin intramuscularly (IM) on day 8. Treatment with LHRH agonist repeats every 12 weeks for 24 weeks.
  Interventions: Drug: bicalutamide; Drug: goserelin; Drug: leuprolide acetate
- Arm II (Experimental): Patients receive androgen ablation as in arm I. Patients receive GVAX prostate cancer vaccine (CG1940 and CG8711) intradermally (ID) on day 1. Beginning on day 1 of week 3, patients receive booster doses of CG1940 and CG8711 ID every 2 weeks for 24 weeks.
  Interventions: Biological: GVAX prostate cancer vaccine; Drug: bicalutamide; Drug: goserelin; Drug: leuprolide acetate

INTERVENTIONS:
Biological: GVAX prostate cancer vaccine — Given intradermally
  Arms: Arm II
Drug: bicalutamide — Given orally
Drug: goserelin — Given intramuscularly
Drug: leuprolide acetate — Given intramuscularly

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Androgen ablation therapy, such as bicalutamide, leuprolide, and goserelin, may lessen the amount of androgens made by the body. Vaccine therapy may help the body build an effective immune response to kill tumor cells. It is not yet known whether androgen ablation therapy is more effective with or without vaccine therapy in treating patients with prostate cancer.

PURPOSE: This randomized phase II trial is studying androgen ablation therapy to see how well it works when given together with or without vaccine therapy in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the median PSA recurrence-free survival of patients with nonmetastatic, biochemically relapsed prostate cancer who respond with a PSA ≤ 0.5 ng/mL when administered a brief (6-month) course of androgen ablation either alone or in combination with GVAX prostate cancer vaccine (CG1940/CG8711) immunotherapy.

Secondary

* To determine the safety of combined treatment with androgen ablation and CG1940/CG8711 immunotherapy in these patients.
* To determine median time to metastatic disease development in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to Gleason score (> 7 vs ≤ 7), PSA doubling time (< 3 months vs 3-9 months vs > 9 months) and prior androgen ablation (yes vs no). Patients are randomized to 1 of 2 treatment arms at a 1 (arm I):2 (arm II) ratio.

* Arm I (androgen-ablation therapy): Patients receive oral bicalutamide once daily on days 1-28. Patients also receive luteinizing hormone-releasing hormone (LHRH) agonist treatment comprising leuprolide acetate or goserelin intramuscularly (IM) on day 8. Treatment with LHRH agonist repeats every 12 weeks for 24 weeks.
* Arm II (androgen-ablation therapy and vaccine): Patients receive androgen ablation as in arm I. Patients also receive GVAX prostate cancer vaccine (CG1940 and CG8711) intradermally (ID) on day 1. Beginning on day 1 of week 3, patients receive booster doses of CG1940 and CG8711 ID every 2 weeks for 24 weeks.

Patients are evaluated on day 1 of week 25 to assess disease. If PSA > 0.5 ng/mL AND there is no evidence of metastatic disease on imaging studies, then patients can be treated at the discretion of the investigator. If PSA ≤ 0.5 ng/mL, and there is no evidence of metastatic disease, then patients are considered responders and continue having PSA evaluated every 4 weeks until PSA relapse.

After completion of study therapy, patients are followed periodically for 5 years and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Biochemically relapsed prostate cancer
* Must have received primary therapy (i.e., radical prostatectomy, definitive radiotherapy, brachytherapy, or cryotherapy)

  * If patient has a rising PSA after radical prostatectomy, salvage radiotherapy must have been offered
* Evidence of biochemical progression as determined by 3 PSA measurements, each higher than the previous value and meeting the following criteria:

  * The second PSA (PSA2) must be obtained at least 8 weeks after the first (PSA1)
  * The third PSA (PSA3) must be obtained at least 2 weeks after the PSA2 and within the past 4 weeks
  * The PSA3 must be > 2.0 ng/mL and ≤ 20 ng/mL
* Must not have received more than 1 course of prior androgen ablation, defined as treatment with a luteinizing hormone-releasing hormone agonist resulting in a castrate testosterone level AND a PSA nadir ≤ 0.1 followed by subsequent withdrawal of androgen ablation and recovery of testosterone to a non-castrate level
* No evidence of metastatic disease on radionuclide bone scan and CT scan performed within the past 8 weeks

  * Retroperitoneal lymphadenectomy ≤ 2 cm is not considered metastatic for purposes of this study

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC > 2,500/mm³
* ANC ≥ 1,500/mm³
* Hemoglobin > 9.0 g/dL
* Platelet count ≥ 100,000/mm³
* Serum creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 60 mL/min
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* PT/INR ≤ 1.3
* Serum testosterone normal
* Fertile patients must use effective contraception
* No active autoimmune disease or history of autoimmune disease requiring treatment with systemic immunosuppression including, but not limited to, any of the following:

  * Inflammatory bowel disease
  * Systemic lupus erythematosus
  * Systemic vasculitis
  * Scleroderma
  * Multiple sclerosis
  * Hemolytic anemia
  * Sjögren syndrome
  * Sarcoidosis
* No known active infection
* No uncontrolled concurrent illness including, but not limited to, any of the following:

  * Systemic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to leuprolide acetate, bicalutamide, or sargramostim (GM-CSF)
* No known sensitivity to materials of bovine origin
* No hypersensitivity to GM-CSF or to any of the other components of CG1940/CG8711, which includes fetal bovine serum, dimethyl sulfoxide (DMSO), and hydroxyethyl starch and may include small amounts of porcine trypsin and DNase

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior and no concurrent systemic corticosteroids

  * Use of inhaled corticosteroids for asthma or chronic obstructive pulmonary disease (COPD) is permitted
* More than 4 weeks since prior and no concurrent chemotherapy or other cancer therapy
* More than 4 weeks since prior and no concurrent use of herbal products (e.g., saw palmetto or PC-SPES)
* At least 4 weeks since prior and no other concurrent investigational agents
* No other concurrent anticancer commercial agents or therapies
* Prior androgen ablation administered concomitantly with primary radiotherapy allowed

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07

PRIMARY OUTCOMES:
Median PSA recurrence-free survival in patients in patients responding to the study treatments

SECONDARY OUTCOMES:
Safety
Effects of 6-month androgen ablation on thymic production of naïve T cells
Median time to metastatic disease development

CONTACTS AND LOCATIONS:
Overall Officials: Charles G. Drake, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Michael A. Carducci, MD — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins